CLINICAL TRIAL: NCT04140851
Title: Effect of Dietary Interventions in Overweight and Obese Patients
Brief Title: Effect of Dietary Interventions on Intestinal Flora and Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuxi Hisky Medical Technology Co Ltd (Industry)
Collaborators: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIIFM-20190701
Record Dates: First submitted 2019-09-29; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Dietary Interventions
Keywords: Dietary Interventions; Intestinal Flora; Metabolism

STUDY DESIGN:
Intervention Model Description: this study enrolled 12 patients with simple overweight or obesity, including 9 males and 3 females. In addition, 20 patients with simple overweight or obesity were randomly selected by comparable age and gender to the control group (excluding criteria), including 11 males and 9 females, and another 20 healthy people were recruited to the healthy control group.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- overweight/obesity diet intervention group (Experimental): Dietary fiber intervention
  Interventions: Dietary Supplement: Dietary fiber intervention
- overweight/obese normal diet group (Placebo Comparator): Normal diet
  Interventions: Dietary Supplement: Normal diet
- healthy control group (No Intervention): Healthy people

INTERVENTIONS:
Dietary Supplement: Dietary fiber intervention — Dietary intervention
  Arms: overweight/obesity diet intervention group
Dietary Supplement: Normal diet — Normal diet
  Arms: overweight/obese normal diet group

SUMMARY:
This study is to explore the effects of dietary intervention on the figure, fatty liver and biochemical indexes; the intestinal flora and metabolomics of the overweight and obese patients.

This study was a clinical control and self-control study (before and after), which enrolled 12 patients with simple overweight or obesity, including 9 males and 3 females. In addition, 20 patients with simple overweight or obesity were randomly selected by comparable age and gender to the control group (excluding criteria), including 11 males and 9 females, and another 20 healthy people were recruited to the healthy control group from the Physical Examination Center, Qilu Hospital of Shandong University.

DETAILED DESCRIPTION:
With the rapid development of China's economy, changes in the residents' living habits and lifestyles, increase in dietary calorie intake, and relative decrease in physical activity, the prevalence of overweight and obesity in China has increased year by year. According to the WGOC diagnostic criteria, the prevalence of overweight and obesity in China was 31.4% and 12.2%, respectively, by 2013. The obesity refers to the chronic metabolic disease caused by the combined action of both genetic and environmental factors. It refers to the weight gain caused by the increase of body fat volume and/or increase of the number of fat cells resulted from the imbalance of energy metabolism, and caloric intake exceeding the calorie consumption. With the prevalence of obesity in the world, the obesity-related chronic diseases have gradually entered the vision of the public, such as non-alcoholic fatty liver disease (NAFLD). The NAFLD refers to the acquired metabolic stress-induced liver injury with diffuse hepatocyte macrobubble fat as clinical pathological syndrome caused by well-defined liver damage factors other than alcohol. It is the most common cause of chronic liver disease in Western countries and also the leading cause for the onset of and death from liver related disease worldwide. The NAFLD is growing rapidly in Asian countries at younger ages. With the increase of obesity rate in the country, the prevalence rate of adult NAFLD in China has also increased rapidly, with the prevalence rate as high as 30% in some areas, and more and more viral hepatitis cases are combined with NAFLD. Therefore, it can be seen that the obesity not only seriously endangers the physical and mental health of the people, but also becomes an important social public health problem that causes disability, affects the quality of life and increases the financial burden of the state. In view of the great harms brought by the obesity, to find a healthy, safe and effective weight loss method has become a public concern and study hotspot. At present, various weight loss treatment methods are available, including dietary control, exercise, and medical and surgical treatment. Each method has its own advantages and disadvantages. The lifestyle intervention based on scientific and rational nutrition therapy combined with exercise is still the safest and most effective weight loss method.

Various methods to lose weight are available so far, such as the dietary control, proper exercise, medical therapy and lately popular gastrointestinal minimally invasive surgery, and each method has its own advantages and disadvantages. The diet drug suppresses the appetite and reduces weight mainly via either central or peripheral means. In the past few decades, many diet drugs have been marketed, such as Phentermine and Sibutramine, etc., but they were soon removed from the market due to limited efficacy, various side effects and addiction, etc. The diet drugs have poor safety and high rebound rate, which also causes serious damage to the body while reducing weight. For the patients with severe obesity, existing surgical procedures, such as volume-limiting surgery, gastric bypass surgery, and the new therapy approved by the FDA in 2014 - vagus nerve block surgery, etc. are really an effective method to lose weight. However, for the patients with overweight and mild obesity, the long-term effects of surgical treatment and postoperative complications prevent them from being used as the preferred method for weight loss. Therefore, the lifestyle intervention based on scientific and rational nutrition therapy and exercise is still the safest and most effective weight loss method so far.

The dietary fiber has been neglected for a period of time for being considered "nutrient-free", and because it is usually the oligosaccharide or polysaccharide that is difficult for digestion and absorption to provide energy to the body. But now more and more studies have shown that dietary fiber is beneficial to intestinal health of human body. The fermented products from dietary fiber, such as short-chain fatty acids (SCFA), can prevent the obesity by regulating appetite, increasing anorexia hormone level and increasing energy consumption, and the addition of soluble dietary fiber to the diet can improve the anthropometric measurements in the overweight or obese patients, and help reduce BMI, the fat, and fasting blood glucose and fasting insulin levels.

The microbial diversity sequencing is the high-throughput sequencing of 16SrDNA hypervariable region of sample bacteria using the new-generation high-throughput sequencing technology (NGS), which is designated to reveal the diversity and structural composition of microbial communities and explore the relationship between the microorganisms and the hosts, so as to provide a theoretical basis for follow-up disease diagnosis and development of microbial resources.

The transient elastography (TE) FibroTouch reflects the degree of hepatic steatosis by measuring the ultrasound attenuation parameters (UAP) of the liver. It is non-invasive, simple, fast, easily operable, repeatable, safe and well tolerable.

The aim of this study is to explore the effects of dietary intervention on the figure, fatty liver and biochemical indexes; the intestinal flora and metabolomics of the overweight and obese patients.

This study was a clinical control and self-control study (before and after), which enrolled 12 patients with simple overweight or obesity, including 9 males and 3 females. In addition, 20 patients with simple overweight or obesity were randomly selected by comparable age and gender to the control group (excluding criteria), including 11 males and 9 females, and another 20 healthy people were recruited to the healthy control group from the Physical Examination Center, Qilu Hospital of Shandong University. Study methods include clinical data collection, FibroTouch detection, stool test, measurement of serum biochemical indicators and analysis of the composition of immune cells in peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* for the overweight/obesity group. Diagnostic criteria for overweight or obesity (basis): The classification standard% for the body mass index of Chinese population [(BMI) = weight (kg)/height square (m^2)] recommended by the Working Group on Obesity of China (WGOC): obesity: BMI ≥ 28 kg/m^2; overweight: 28 kg/m^2 > BMI ≥ 24 kg/m^2; normal weight: 24 kg/m^2 > BMI ≥18.5 kg/m^2; underweight: BMI < 18.5 kg/m^2;
* The subjects had not received weight loss treatment such as being on diet, diet drugs or surgery 6 months before the enrollment;
* The subjects signed the informed consent form, and were able and willing to adhere to low-carbohydrate diet and receive regular call and outpatient follow-up;

Exclusion Criteria:

* pregnant women, lactating women or women planning to get pregnant;
* the obesity caused by endocrine system and central nervous system diseases or drugs, type 2 diabetes, autoimmune diseases and other endocrine systemic diseases;
* history of acute or chronic infection, surgery or trauma, or history of malignant tumor;
* severe liver and kidney dysfunction (transaminase > 2.5 times of normal upper limit); creatinine: male ≥ 133 μmol/L; female ≥ 124 μmol/L;
* the patients with severe heart, brain or peripheral vascular diseases;
* Those unable to cooperate with the observer for various reasons.

The subjects withdrew from the criteria:

* being unable to continue the intervention due to other reasons or diseases during the treatment;
* being unsatisfied with the improvement in the symptoms during the treatment and requiring to stop the trial;
* having serious adverse events or adverse reactions, and the investigator considers it is necessary for the subject to terminate the trial from the medical perspective.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
The value of Ultrasound Attentunation Parameter in the overweight and obese patients | 3 months
  Liver is detected by FibroTouch to get UAP showing liver steatosis in obesity
The serological indexes in the overweight and obese patients | 3 months
  Serological testing gets a series of serological indicator, such as AST/ALT (U/L)

SECONDARY OUTCOMES:
The composition of immune cells in peripheral blood of the overweight and obese patients | 3 months
  Perform immune cell sorting by flow cytometry, and analyze the proportion of various immune cells; analyze the proportion of 22 kinds of immune cells
The composition of intestinal flora of the overweight and obese patients | 3 months
  Stool test gets the composition of intestinal flora.

CONTACTS AND LOCATIONS:
Overall Officials: Fuqiang Liu, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Liu Fuqiang, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Zhao L, Zhang F, Ding X, Wu G, Lam YY, Wang X, Fu H, Xue X, Lu C, Ma J, Yu L, Xu C, Ren Z, Xu Y, Xu S, Shen H, Zhu X, Shi Y, Shen Q, Dong W, Liu R, Ling Y, Zeng Y, Wang X, Zhang Q, Wang J, Wang L, Wu Y, Zeng B, Wei H, Zhang M, Peng Y, Zhang C. Gut bacteria selectively promoted by dietary fibers alleviate type 2 diabetes. Science. 2018 Mar 9;359(6380):1151-1156. doi: 10.1126/science.aao5774. PMID 29590046
- [Background] Canfora EE, Meex RCR, Venema K, Blaak EE. Gut microbial metabolites in obesity, NAFLD and T2DM. Nat Rev Endocrinol. 2019 May;15(5):261-273. doi: 10.1038/s41574-019-0156-z. PMID 30670819
- [Background] Thompson SV, Hannon BA, An R, Holscher HD. Effects of isolated soluble fiber supplementation on body weight, glycemia, and insulinemia in adults with overweight and obesity: a systematic review and meta-analysis of randomized controlled trials. Am J Clin Nutr. 2017 Dec;106(6):1514-1528. doi: 10.3945/ajcn.117.163246. Epub 2017 Nov 1. PMID 29092878
- [Background] Zhuang Xiaofang, et al. Evaluation of the performance of transient elastography in the diagnosis of nonalcoholic fatty liver disease. Journal of Clinical Hepatology, 33(12): 2366-2371.
- [Background] Leng Xuejun. et al. Evaluation and comparison with FibroTouch® the degree of liver fibrosis in the patients with nonalcoholic fatty liver disease of different BMI levels. Journal of Clinical Hepatology, 34(9): 1891-1895.